CLINICAL TRIAL: NCT07209150
Title: Randomized Controlled Trial of 3 vs 7 Days for Perioperative Antibiotic Prophylaxis for Patients With an Indwelling Catheter Prior to Holmium Laser Enucleation of the Prostate
Brief Title: Randomized Controlled Trial of Different Antibiotic Duration Prior to Prostate Enucleation Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025HoLEP_periopabx
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: BPH With Urinary Obstruction; Antibiotic Prophylaxis
Keywords: bph; urinary retention; antibiotic prophylaxis
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Retention | interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Intervention Model Description: Patients who are eligible to undergo HoLEP and have an indwelling urinary catheter or perform CIC will be randomized to different durations of peri-operative antibiotic prophylaxis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 day prophylaxis (Experimental): 3 days of perioperative culture directed antibiotic prophylaxis will be prescribed to this group (to start 1 day prior to surgery). macrobid if preoperative culture is negative
  Interventions: Drug: antibiotic prophylaxis
- 7 day prophylaxis (Other): 7 days of perioperative culture directed antibiotic prophylaxis will be prescribed to this group (to start 4 day prior to surgery). macrobid if preoperative culture is negative
  Interventions: Drug: antibiotic prophylaxis

INTERVENTIONS:
Drug: antibiotic prophylaxis — we will compare varying durations of antibiotic prophylaxis prior to prostate enucleation surgery

SUMMARY:
To compare the risk of infectious complications (UTI, pyelonephritis, sepsis, hospital admission, ED visits) for patients with an indwelling urinary catheter (urethral or suprapubic) or CIC receiving 3 or 7 days of peri-operative antibiotic prophylaxis at time of Holmium Laser Enucleation of the Prostate

ELIGIBILITY:
Inclusion Criteria:

* 1. Candidate for HoLEP surgery 2. Must be 18 years or older. 3. The patient must be able to understand and willing to provide informed consent as described in this study protocol.

Exclusion Criteria:

* 1. Under the age of 18 2. Refuse to provide informed consent 3. Anticipated need for perineal urethrostomy 4. History of multi-drug resistant organism on urine culture that is not susceptible to any oral agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Infectious complications | 0-90 days postoperatively
  UTI, pyelonephritis, sepsis, hospital admission, ED visits

SECONDARY OUTCOMES:
healthcare utilization | 0-90days
  hospital admission or ED visits occurring post HoLEP

IPD SHARING:
Plan to Share IPD: No